CLINICAL TRIAL: NCT00849069
Title: An Observer-blind, Safety Study of GSK Biologicals' Haemophilus Influenzae and Streptococcus Pneumoniae Candidate Vaccine in Adults.
Brief Title: Study to Assess the Safety of a New GSK Biologicals' GSK2231395A Candidate Vaccine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study has been stopped for logistic reasons not related to the safety or efficacy of the vaccine.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 112350
Record Dates: First submitted 2009-02-19; First posted 2009-02-23 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Haemophilus Influenzae; Streptococcus Pneumoniae
Keywords: Streptococcus pneumoniae; Vaccine; Non-typable Haemophilus influenza; Adults and Elderly Adults
MeSH Terms: conditions — Haemophilus Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: GSK2231395A
- Group B (Active Comparator)
  Interventions: Biological: TwinrixTM

INTERVENTIONS:
Biological: GSK2231395A — 3 doses intramuscular injections
  Arms: Group A
Biological: TwinrixTM — 3 doses intramuscular injections
  Arms: Group B

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity and immunogenicity of GSK2231395A candidate vaccine in adults and elderly adults with chronic obstructive pulmonary disease. Subjects will be vaccinated 3 times with an interval of respectively 2 and 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, 40 and 80 years of age, inclusive, at the time of consent.
* Written informed consent obtained from the subject.
* Subject has a confirmed history of chronic obstructive pulmonary disease exacerbations, including multiple exacerbations in the 24 months prior to Screening
* Subject has a baseline chest X-ray obtained while untreated/off systemic corticosteroids for at least 30 days duration
* Subject is able to perform baseline pre- and post-bronchodilator pulmonary function tests while untreated/off systemic corticosteroids for at least 30 days duration and not participating in a pulmonary rehabilitation program.
* If the subject is female, and of childbearing potential, she agrees to use acceptable contraception and not become pregnant for the duration of the study.

Exclusion Criteria:

* Is established by a screening pulmonary function test as having mild chronic obstructive pulmonary disease
* Is established by both a screening PFT and clinical history as having very severe chronic obstructive pulmonary disease
* Is diagnosed with a respiratory disorder other than chronic obstructive pulmonary disease
* Has a primary diagnosis of asthma.
* Is prescribed/receiving systemic antibiotics in the last 30 days.
* Is prescribed/receiving systemic corticosteroids in the last 30 days.
* Has chronic administration of immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccine dose.
* Is undergoing, planning to undergo, or has undergone in the last 6 months a pulmonary rehabilitation program.
* Has undergone, or planning to undergo, lung transplantation and/or lung volume reduction.
* Has chest x-ray indicating an acute pulmonary disease requiring therapy or that might interfere with the study, such as CAP, tuberculosis, or lung cancer
* Has had pneumonia within 3 months prior to first vaccination.
* Is receiving regular long-term oxygen therapy.
* Has a known diagnosis of α-1 antitrypsin deficiency.
* Has a known or suspected hypersensitivity/reaction to any components of the candidate vaccine, the comparator vaccine (Twinrix® Adult or any ingredient), and/or the bronchodilator used in the study procedures.
* Has been previously vaccinated for Hepatitis A and/or B. As a portion of the subjects will be randomized to receive Twinrix® Adult comparator, it is important that all subjects qualify to receive Twinrix® Adult.
* Is using any investigational or non-registered product (drug or vaccine) other than the study vaccine, within 30 days preceding the first dose of study vaccine, or planned use during the study period, or participation to another pharmaceutical/vaccine study.
* Has administered, or is planning administration, of any vaccine not foreseen by the study protocol within 30 days of the first dose of vaccines.
* Has administration of immunoglobulins and/or any blood products within the 3 months prior to first vaccination.
* Has any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* Has significant disease, in the opinion of the investigator, likely to interfere with the study and/or likely to cause death within the study duration.
* Has acute cardiac insufficiency.
* Has inflammatory processes such as known chronic active infections (e.g. Hepatitis B, Hepatitis C).
* Has past or current malignancies and lymphoproliferative disorders.
* Has clinically significant hematological or biochemical abnormalities as per the judgment of the investigator.
* Has acute disease at the time of vaccination.
* Is a pregnant or lactating female.
* Is female and is planning to become pregnant or planning to discontinue contraceptive precautions.
* Has, in the opinion of the investigator, evidence of alcohol or drug abuse.
* Has other conditions that the principal investigator judges may interfere with study findings.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-03-12 (Actual); Primary Completion 2009-04-07 (Actual); Study Completion 2009-04-07 (Actual)

PRIMARY OUTCOMES:
Occurrence, intensity and relationship of adverse events after each vaccine dose. | Defined period in function of the measured parameter
Occurrence of any vaccine-related serious adverse events | Throughout the study
Occurrence of any adverse event of specific interest | Throughout the study

SECONDARY OUTCOMES:
Evaluation of the disease progression of subjects receiving the candidate vaccine versus subjects receiving the comparator vaccine. | Defined time points in function of the measured parameter
Evaluation of antibody responses against candidate vaccine antigens. | Defined time points in function of the measured parameter
Evaluation of the clinical outcomes of subjects receiving the candidate vaccine versus subjects receiving the comparator vaccine. | Defined time points in function of the measured parameter

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Halifax, Nova Scotia, Canada